CLINICAL TRIAL: NCT06007222
Title: Non-antithrombotic Therapy After Transcatheter Aortic Valve Implantation Trial
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: OCEAN-SHD Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAPT trial
Record Dates: First submitted 2023-08-08; First posted 2023-08-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Aortic Stenosis; TAVI(Transcatheter Aortic Valve Implantation); Aspirin; DAPT(Dual Antiplatelet Therapy); SAPT(Single Antiplatelet Therapy)
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspirin group (Active Comparator): Aspirin 100mg will be started within 24 hours after randomization, and continued aspirin 100mg/day the end of the study period.
  Interventions: Drug: Aspirin group
- Non-antithrombotic group (Experimental): No antithrombotic agents will be administered after randomization until the end of the study period.
  Interventions: Drug: Non-antithrombotic group

INTERVENTIONS:
Drug: Aspirin group — Aspirin 100mg will be started within 24 hours after randomization, and continued aspirin 100mg/day the end of the study period.
  Arms: Aspirin group
Drug: Non-antithrombotic group — No antithrombotic agents will be administered after randomization until the end of the study period.
  Arms: Non-antithrombotic group

SUMMARY:
Aspirin group: Aspirin 100mg will be started within 24 hours after randomization, and continued aspirin 100mg/day the end of the study period.

Non-antithrombotic group: No antithrombotic agents will be administered after randomization until the end of the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent transfemoral TAVI for aortic stenosis
2. Patients aged 20 years or older at the time of informed consent
3. Patients who have a thorough understanding of the subject of the study and who have agreed in writing to participate in the study

Exclusion Criteria:

1. Those with perioperative complications at the time of TAVI (conversion to open heart surgery, coronary artery occlusion, annulus rupture, cardiac tamponade, vascular dissection, cerebral infarction/cerebral hemorrhage, new atrial fibrillation, new atrioventricular block)
2. Individuals requiring antiplatelet agents for reasons other than TAVI (history of myocardial infraction, history of PCI（Percutaneous Coronary Intervention）, history of EVT（EndoVascular Treatment）, history of cerebral infraction and transient ischaemic stroke, with significant coronary artery narrowing, with high-grade carotid artery narrowing, and others judged as requiring antiplatelet therapy by the chief researcher or a sub-investigator)
3. Patients requiring oral anticoagulants (patients with atrial fibrillation, history of pulmonary embolism or deep venous thrombosis, and other patients who are deemed to require anticoagulation therapy by the investigator or coinvestigator)
4. Patients with eGFR（estimated Glomerular Filtration Rate） <30 and patients on hemodialysis/peritoneal dialysis.
5. Patients with a history of valve replacement in the heart valves.
6. Patients who are pregnant, have childbearing potential, wish to become pregnant, or are breastfeeding.
7. Patients who have a concomitant medical illness associated with expected survival less than one year.
8. Patients who have the contraindications for aspirin.
9. Patients with a diagnosis of severe allergy to aspirin or a history of hypersensitivity.
10. Patients requiring a legally acceptable representative, patients unable to obtain written informed consent, or patients unable to understand the outline or purpose of the study.
11. Other patients for whom the principal investigator or the coinvestigator judges the participation in the study inappropriate.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | minimum 2 years, maximum 3 years of follow-up
  Composite endpoint consisting of all-cause deaths, myocardial infarction, stroke from any cause and bleeding from randomization to end of study
  The outcomes of this study will comply with the Valve Academic Research Consortium 3 (VARC 3). VARC 3 Type 1, Type 2, Type 3, and Type 4 bleeding are all included as bleeding. In this study, the study subjects will be randomized after it has been confirmed that there were no perioperative complications, so it is essentially assumed that there will be no procedure-related bleeding.
  Surviving subjects for whom the event does not occur will be censored as of the date the study treatment is discontinued or as of the last confirmed date of survival.

SECONDARY OUTCOMES:
Key Secondary endpoint | minimum 1 year, maximum 3 years of follow-up
  Bleeding Events from Randomization to Study End. Cardiovascular adverse events from randomization until the end of the study (composite endpoint comprised of cardiovascular death, myocardial infarction, or CVA).
  The definition of censoring for survival time analysis is the same as that used for the primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Yosuke Sawa, Study Director — EPS Corporation
Locations (1):
- Keio University Hospital, Shinjuku, Tokyo, Japan